CLINICAL TRIAL: NCT03890042
Title: Dienogest Versus a Low-dose Combined Oral Contraceptive for Treatment of Adenomyotic Uteri
Brief Title: Dienogest for Treatment of Adenomyotic Uteri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAD
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Femovan; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dienogest group (Active Comparator)
  Interventions: Drug: Dienogest group; Radiation: Ultrasound; Other: visual analogue scale
- Gynera group (Active Comparator)
  Interventions: Drug: Gestodene-Ethinyl Estradiol; Radiation: Ultrasound; Other: visual analogue scale

INTERVENTIONS:
Drug: Dienogest group — VISANNE 2MG Tablet once daily
  Arms: Dienogest group
Drug: Gestodene-Ethinyl Estradiol — Gynera tablet once daily
  Arms: Gynera group
Radiation: Ultrasound — ultrasound assessment of uterine volume
Other: visual analogue scale — visual analogue scale for assessment of pain

SUMMARY:
Adenomyosis is a common disease in women aged 40-50 years. It associates with dysmenorrhea and menorrhagia. Hysterectomy was considered the main treatment that could definitively cure this disease. Other treatment options are increasingly offered, including hormonal suppression with gonadotropin-releasing hormone agonists or danazol and endometrial ablation. However, deep adenomyosis responds weakly to the above treatment options, which are commonly not considered for long-term management because of the associated side effects.

Dienogest is a progestin medication which is used in birth control pills and in the treatment of endometriosis and adenomyosis. Low-dose combined oral contraceptive (COC) pills have been widely used as the primary treatment for menorrhagia. COCs can also be used to induce endometrial atrophy and to decrease endometrial prostaglandin production, which can consequently improve menorrhagia and dysmenorrhea that are associated with adenomyosis

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-40 years
* Women with ultrasonographic evidence of adenomyosis
* Woman complains of vaginal bleeding or pelvic pain related to adenomyosis

Exclusion Criteria:

* Women with a history of malignancy or histological evidence of endometrial hyperplasia
* any adnexal abnormality on ultrasound
* undiagnosed vaginal
* contraindication to receive Vissane or gynera .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Number of women who will improved from the pelvic pain measured by visual analogue scale | 6 months

SECONDARY OUTCOMES:
Uterine volume (cm 3 ) measure by ultrasound | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

REFERENCES:
- [Derived] Hassanin AI, Youssef AA, Yousef AM, Ali MK. Comparison of dienogest versus combined oral contraceptive pills in the treatment of women with adenomyosis: A randomized clinical trial. Int J Gynaecol Obstet. 2021 Aug;154(2):263-269. doi: 10.1002/ijgo.13600. Epub 2021 Feb 11. PMID 33454995